CLINICAL TRIAL: NCT02414373
Title: Effects of Thoracic Epidural Administered Ropivacaine Versus Bupivacaine on Lower Urinary Tract Function: A Randomized, Controlled Study
Brief Title: Effects of Thoracic Epidural Administered Ropivacaine Versus Bupivacaine on Bladder Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390/14
Record Dates: First submitted 2015-03-26; First posted 2015-04-10 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Post Operative Urinary Retention
Keywords: urination; analgesia, epidural; local anesthetics
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine 2mg/ml (ROPIVACAIN Sintetica 2 mg/ml ™, Sintetica-Bioren, Couvet, Schweiz)
  Interventions: Drug: Ropivacaine 2mg/ml; Device: 6 French transurethral dual channel catheter (Gaeltec, Dunvegan, Scotland); Device: 14 French rectal balloon catheter (Gaeltec, Dunvegan, Scotland)
- Bupivacaine (Active Comparator): Bupivicaine 1.25mg/ml (BUPIVACAIN Sintetica 0.125 % ™ (Bupivacain 1,25 mg/ml), Sintetica-Bioren, Couvet, Schweiz)
  Interventions: Drug: Bupivacaine; Device: 6 French transurethral dual channel catheter (Gaeltec, Dunvegan, Scotland); Device: 14 French rectal balloon catheter (Gaeltec, Dunvegan, Scotland)

INTERVENTIONS:
Drug: Ropivacaine 2mg/ml — local anesthetics, which will epidurally administered
  Arms: Ropivacaine
Drug: Bupivacaine — local anesthetics, which will epidurally administered
  Arms: Bupivacaine
Device: 6 French transurethral dual channel catheter (Gaeltec, Dunvegan, Scotland)
Device: 14 French rectal balloon catheter (Gaeltec, Dunvegan, Scotland)

SUMMARY:
Acute urinary retention is one of the most common complications after surgery and anesthesia. Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Under the influence of epidural analgesia, patients may not feel the sensation of bladder filling, which can result in urinary retention and bladder overdistension. Overfilling of the bladder can stretch and in some cases permanently damage the detrusor muscle. Because epidural anesthesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Thoracic epidural analgesia with bupivacaine significantly inhibits the detrusor muscle during voiding, resulting in clinically relevant post void residuals which required monitoring or transurethral catheterisation. This bladder muscle inhibition is comparable to a motor blockade. The epidural administration of ropivacaine during labour results in a clinically relevant reduction of motor blocks.

The hypothesis is that thoracic epidural analgesia with the local anesthetics ropivacaine leads to less significant changes in bladder function than bupivacaine as a control group, in patients undergoing lumbotomy incision for renal surgery.

DETAILED DESCRIPTION:
Background

Acute urinary retention is one of the most common complications after surgery and anesthesia. It can occur in patients of both sexes and all age groups and after all types of surgical procedures. It is linked to several factors including increased intravenous fluids, postoperative pain and type of anaesthesia.

Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord and coordination between them occurs in the pontine tegmentum of the caudal brain stem. Motorneurons innervating the external urethral sphincter are located in the nucleus of Onuf, extending from segment S1 to S3. The detrusor smooth muscle is innervated by parasympathetic fibers, which reside in the sacral intermediolateral cell group and are located in S2-4. Sympathetic fibers innervating the bladder and urethra play an important role in promoting continence and are located in the intermediolateral cell group of the lumbar cord (L1-L4). Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2 and the majority are thin myelinated or unmyelinated.

There are few studies on the urodynamic effects of various anaesthetic agents, which mainly focused on lumbar epidural anaesthesia. Under the influence of epidural analgesia, patients may not feel the sensation of bladder filling, which can result in urinary retention and bladder overdistension. Overfilling of the bladder can stretch and in some cases permanently damage the detrusor muscle.

Because epidural anesthesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Based on knowledge of the bladder innervations, it can be assumed that epidural analgesia within segments T4-6 to T10-12 has no or minimal influences on lower urinary tract function.

In a previous study, the investigators found, against their expectations, that thoracic epidural analgesia (TEA) with bupivacaine significantly inhibits the detrusor muscle during voiding, resulting in clinically relevant post void residuals which required monitoring or transurethral catheterisation 11. This detrusor inhibition is comparable to a motor blockade.

In addition, it is known that the epidural administration of ropivacaine during labour results in a clinically relevant reduction of motor blocks. However, the analgesic potency of ropivacaine is approximately 60% that of bupivacaine.

Objective

The main objectives of this investigator initiated trial are:

* To analyse if a TEA with the local anesthetics ropivacaine leads to less detrusor atony and thus resulting to lower incidence of postvoid residual urine volume resulting in postoperative urinary retention.
* To compare urodynamic parameters (storage and voiding phases) during TEA with ropivacaine versus bupivacaine.

Methods

Assessments of bladder function:

International Prostate Symptom Score (IPSS) will be used for assessment of lower urinary tract symptoms preoperatively.

Urodynamic investigations will be performed: The first investigation will be done as baseline data before attempted surgery.

Urodynamic investigations will be performed according to good urodynamic practice. After placement of a 6 French transurethral dual channel catheter and a 14 French rectal balloon catheter (Gaeltec, Dunvegan, Scotland), the bladder will be filled at a rate of 25 to 50 ml/min with Ringer's lactate solution at room temperature. Parameters of both the storage phase (maximum cystometric capacity, bladder compliance) and voiding phase (detrusor pressure at maximum flow rate (PdetQmax), maximum flow rate (Qmax) and PVR will be recorded. All methods, definitions and units will be in accordance with the standards recommended by the International Continence Society.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Kidney surgery
* Thoracic epidural analgesia

Exclusion Criteria

* Contraindications to epidural analgesia or refusal
* Preoperative postvoid residual urine volume > 100ml
* International Prostate Symptom Score (IPSS) > 7
* Pregnancy (pregnancy test in all women who are not in menopause, exclusion for surgery per se)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Post void residual urine volume: Change between postvoid residual urine volume before surgery versus during thoracic epidural analgesia for postoperative analgesia | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)

SECONDARY OUTCOMES:
Bladder volume at first desire to void (mL) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Maximum cystometric capacity (mL) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Bladder compliance (mL/cmH2O) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Urethral pressure profile (cmH2O) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Maximum detrusor pressure (cmH2O) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Detrusor pressure at maximum flow rate(cmH2O) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.
Maximum flow rate (mL/sec) | before surgery/TEA (baseline), during TEA (expected to be on average ca. 5 days)
  Change of the parameters of the storage and voiding phases from baseline (preoperative) to postoperative day 2 or 3, depending on patient's mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wuethrich, MD, Principal Investigator — Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, 3010 Bern
Locations (1):
- Patrick Wuethrich, Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, Bern, Canton of Bern, Switzerland